CLINICAL TRIAL: NCT05482152
Title: Effect Van Preklinische Nurse-led Neuroscience Pijneducatie op de Attituden Ten Opzichte Van Chronische Pijn en de patiënttevredenheid in Een Universitair Pijncentrum: Een Monocentrische RCT
Brief Title: Nurse-led Pain Education Clinical Trial in Chronic Pain Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Filip Haegdorens, Principal Investigator, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: S65953
Record Dates: First submitted 2022-01-13; First posted 2022-08-01 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard physician led care (No Intervention): Consultation by physician (pain specialist)
- Nurse-led care (Experimental): Preclinical nurse-led consultation and standard care by physician (pain specialist)
  Interventions: Behavioral: Nurse-led care by a nurse specialist in pain

INTERVENTIONS:
Behavioral: Nurse-led care by a nurse specialist in pain — A nurse pain specialist consultation in patients in the experimental arm before they receive standard care by a physician.
  Arms: Nurse-led care

SUMMARY:
Chronic pain is a multidimensional problem that consequently requires interventions on multiple levels. Pain education by physicians is one of the interventions that shows promising results in patient reported outcomes. It is however unclear if nurse-led chronic pain education could be equally effective on pain attitude and behavior in chronic pain patients. The aim of this clinical trial is to investigate the effects of a nurse-led consultation with chronic pain patients on pain attitude and patient satisfaction compared with regular care without nurse specialist intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old
* dutch speaking
* first time consultation

Exclusion Criteria:

* Palliative care patients
* Patients with dementia diagnosis
* Urgent referral to the pain clinic by other physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Patient attitude on chronic pain | Up to 10 months
  Pain Solutions Questionnaire (PaSol)

SECONDARY OUTCOMES:
Patient satisfaction | Up to 10 months
  Core questionnaire for the assessment of patient satisfaction in academic hospitals (COPS)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Morlion, MD PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZLeuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided